CLINICAL TRIAL: NCT01890148
Title: An Explorative Investigation to Study the Relationship and Distribution of Neutrophils in Bronchial Mucosal Tissue, Induced Sputum and Blood After Administration of 45 mg BD AZD 5069 for 4 Weeks to Patients With Moderate Persistent Neutrophilic Asthma
Brief Title: Distribution of Neutrophils in Bronchial Mucosal Tissue in Asthma Patients Before and After 4 Weeks Treatment With AZD 5069
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: D3551C00003
Record Dates: First submitted 2013-06-17; First posted 2013-07-01 (Estimated); Results first posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-01

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — N-(2-(2,3-difluoro-6-benzylthio)-6-(3,4-dihydroxybutan-2-yloxy)pyrimidin-4-yl)azetidine-1-sulfonamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): oral BD administration of 45 mg AZD5069
  Interventions: Drug: AZD5069

INTERVENTIONS:
Drug: AZD5069 — oral BD administration of 45 mg AZD5069

SUMMARY:
Distribution of neutrophils in bronchial mucosal tissue in asthma patients before and after 4 wk treatment with AZD 5069

DETAILED DESCRIPTION:
The purpose is to investigate the bronchial tissue neutrophil counts and distribution in asthma patients after 4 week oral treatment with AZD 5069

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients of Caucasian origin, aged between 18 to 65 years, inclusive, at the time informed consent is obtained.
2. Physician based (according to GINA 2011) diagnosis of asthma for at least 6 months prior to the date informed consent is obtained and confirmed by 1 of the detailed respiratory criteria stated in the CSP
3. Morning prebronchodilator (ie, after abstinence from short-acting and long-acting ß-agonist treatment for ≥ 6 and ≥ 12 hours, respectively) FEV1 of ≥70% of predicted normal (PN) for age, sex and height at enrolment
4. Increased number of neutrophils in induced sputum samples at baseline, with a relative neutrophil count of ≥ 50% of total sputum cell count
5. Physician prescribed daily use of medium or high dose ICS (≥ fluticasone 250 μg to ≤ 1.000 µg or the equivalent daily, as defined in GINA 2011; see CSP Appendix E) plus LABA.

Exclusion Criteria:

1. History of clinically relevant allergies or idiosyncrasies to AZD5069 or other investigational CXCR2 antagonists, or any inactive ingredient(s) of the IMP, or tool-substances (eg, salbutamol, local anaesthetics) used for the purpose of this study
2. History of severe asthma exacerbation requiring hospitalization within the last 12 months before screening.
3. Asthma exacerbation requiring a treatment course of systemic (ie, oral or parenteral) corticosteroids within the 3 months before screening or ≥ 3 courses within the last 12 months before screening.
4. Moderate to severe airflow limitation (FEV1 <70% PN)
5. Any chronic lower respiratory disease other than asthma (see CSP for details) that, as judged by the Investigator or Medical Monitor, would interfere with the evaluation of the IMP or interpretation of patient safety or study results.

   -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kai Richter, MSD, Study Director — Astrazeneca Sweden; Klaus F Rabe, MD, Principal Investigator — Lung Clinic Grosshansdorf Germany
Locations (1):
- Research Site, Großhansdorf, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirteen patients were screened; 8 patients were screening failures, 5 patients were enrolled in the study and received treatment with AZD5069.
  First patient enrolled: 11 March 2014. Last patient completed: 18 August 2014.
Groups:
- AZD5069: AZD5069 45mg oral twice daily (BID)
Period: Overall Study
Arm/Group | AZD5069
Started | 5
Completed | 4
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | AZD5069
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Summary for Change From Baseline of Mean Global Semi-quantitative Score Values for Neutrophils in Bronchial Biopsies
Description: Change from baseline reflects the Week 4 value minus the baseline value. Baseline value is Day-14 measurement.
  For semi-quantitative scores, 1= few number of Neutrophils, 2= moderate number of Neutrophils, 3= abundant of Neutrophils. For this end point the reduction in mean of semi-quantitative (arbitrary) scores indicates better result, i.e. lower numbers of Neutrophils.
  The scores given for the biopsies taken at screening and end of treatment is the mean global semi-quantitative scores for the three compartments intraepithelial, subepithelial and submucosal.
Time Frame: Baseline and Week 4
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AZD5069
Number analyzed (Participants) | 4
Units on a scale | -1.21 (0.54)

2. Primary Outcome: Summary for Change From Baseline Neutrophils in Sputum
Description: Change from Baseline reflects the Day 8, Day22 and Day29 minus the baseline value.
Time Frame: Baseline, Day 8, Day 22 and Day29
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | AZD5069
Number analyzed (Participants) | 4
10^9 cells/L
  Day 8 | -4.294 (3.062)
  Day 22 | -6.670 (3.751)
  Day 29 | -3.849 (1.861)

3. Primary Outcome: Summary for Change From Baseline Neutrophil Cell Counts in Blood
Description: Change from Baseline reflects the Day 2, Day 8, Day 15, Day 22, Day29 and Day 34 minus the baseline value
Time Frame: Baseline, Day 2, Day 8, Day 15, Day 22, Day29 and Day 34
Population: PD Analysis
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | AZD5069
Number analyzed (Participants) | 4
10^9 cells/L
  Day 2 | -2.517 (0.420)
  Day 8 | -1.494 (0.559)
  Day 15 | -1.985 (0.425)
  Day 22 | -1.658 (0.237)
  Day 29 | -1.178 (1.375)
  Day 34 | -0.306 (0.200)

4. Secondary Outcome: Summary for Change From Baseline for IL-8 by Type of Sample
Description: Change from baseline reflects the Day 29 value minus the baseline value.
Time Frame: Baseline and Day 29
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | AZD5069
Number analyzed (Participants) | 4
pg/ml
  IL-8 in Serum | 46.88 (34.13)
  IL-8 in Sputum | 5780.75 (3763.83)

5. Secondary Outcome: Summary for Change From Baseline for GRO-alpha by Type of Sample
Description: Change from baseline reflects the Day 29 value minus the baseline value.
Time Frame: Baseline and Day 29
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | AZD5069
Number analyzed (Participants) | 4
pg/ml
  GRO-alpha in Serum | 179.75 (98.20)
  GRO-alpha in Sputum | 7352.50 (22373.99)

6. Secondary Outcome: Summary for Change From Baseline for MMP-9 by Type of Sample
Description: Change from baseline reflects the Day 29 value minus the baseline value.
Time Frame: Baseline and Day 29
Population: PD analysis
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | AZD5069
Number analyzed (Participants) | 4
ng/ml
  MMP-9 in Serum | -157.75 (289.76)
  MMP-9 in Sputum | -80.75 (178.55)

7. Secondary Outcome: Summary Statistics for AUC0-4hrs on Day 29/ Visit T7 (PK Analysis Set)
Description: Summary statistics including geometric mean and standard error for AUC0-4hrs on Day 29/ Visit T7 (PK analysis set).
  Plasma concentration data beyond 0.5 hrs post dose at Day 29 were missing for one patient. For this patient only Cmin value was reported and the AUC0-4hrs and Cmax values were not reported.
Time Frame: At 0, 0.5, 1, 1.5, 2, 2.5, 3, 4 hours post dose on Day 29 (Visit T7)
Measure: Geometric Mean (Standard Error); unit: h*nmol/L
Arm/Group | AZD5069
Number analyzed (Participants) | 3
h*nmol/L | 8571.72 (2421.99)

8. Secondary Outcome: Summary Statistics for Cmin on Day 29/ Visit T7 (PK Analysis Set)
Description: Summary statistics including geometric mean and standard error for Cmin on Day 29/ Visit T7 (PK analysis set).
  Plasma concentration data beyond 0.5 hrs post dose at Day 29 were missing for one patient. For this patient only Cmin value was reported and the AUC0-4hrs and Cmax values were not reported.
Time Frame: At 0, 0.5, 1, 1.5, 2, 2.5, 3, 4 hours post dose on Day 29 (Visit T7)
Measure: Geometric Mean (Standard Error); unit: nmol/L
Arm/Group | AZD5069
Number analyzed (Participants) | 4
nmol/L | 466.92 (272.3)

9. Secondary Outcome: Summary Statistics for Cmax on Day 29/ Visit T7 (PK Analysis Set)
Description: Summary statistics including geometric mean and standard error for Cmax on Day 29/ Visit T7 (PK analysis set).
  Plasma concentration data beyond 0.5 hrs post dose at Day 29 were missing for one patient. For this patient only Cmin value was reported and the AUC0-4hrs and Cmax values were not reported.
Time Frame: At 0, 0.5, 1, 1.5, 2, 2.5, 3, 4 hours post dose on Day 29 (Visit T7)
Measure: Geometric Mean (Standard Error); unit: nmol/L
Arm/Group | AZD5069
Number analyzed (Participants) | 3
nmol/L | 3565.76 (762.84)

10. Secondary Outcome: Number of Adverse Events
Description: Summary of number of adverse events (safety set)
Time Frame: Up to 40 days
Measure: Number; unit: adverse events
Arm/Group | AZD5069
Number analyzed (Participants) | 5
adverse events
  Total number of unique AEs | 10
  Total number of AEs | 11
  Total number of SAEs | 0

11. Secondary Outcome: Number of Participants With Adverse Events
Description: Summary of number of participants with adverse events (safety set)
Time Frame: Up to 40 days
Measure: Number; unit: Participants
Arm/Group | AZD5069
Number analyzed (Participants) | 5
Participants
  Total number of subjects with at least one AE | 4
  Number of subjects withdrawn from study due to AE | 1

12. Secondary Outcome: Summary Statistics for Patient Diary Variables (Day Time)
Description: Summary statistics for patient diary variable, observations with no asthma symptoms (day time), by period (safety set).
  The screening period was Day -14 to -1. Period 1 was the first half of treatment period, Day 1 to daytime record Day 15. Period 2 was the second half of treatment period, night-time record Day 15 to night-time record Day 29+1.
  One participant left the study on day 2, due to adverse event.
Time Frame: Up to 44 days
Measure: Number; unit: Observations
Units Other Than Participants: Observation
Arm/Group | AZD5069
Number analyzed (Participants) | 5
Number analyzed (Observation) | 197
Observations
  Obs. with No asthma symptoms (Screening; n=55) | 6
  Obs. with No asthma symptoms (Period1; n=71) | 7
  Obs. with No asthma symptoms (Period2; n=71) | 7

13. Secondary Outcome: Summary Statistics for Patient Diary Variables (Night Time)
Description: Summary statistics for patient diary variable, observations with no asthma symptoms (night time), by period (safety set).
  The screening period was Day -14 to -1. Period 1 was the first half of treatment period, Day 1 to daytime record Day 15. Period 2 was the second half of treatment period, night-time record Day 15 to night-time record Day 29+1.
  One participant left the study on day 2, due to adverse event.
Time Frame: Up to 44 days
Measure: Number; unit: Observations
Units Other Than Participants: observations
Arm/Group | AZD5069
Number analyzed (Participants) | 5
Number analyzed (observations) | 191
Observations
  Obs. with No asthma symptoms (Screening; n=52) | 9
  Obs. with No asthma symptoms (Period1; n=69) | 2
  Obs. with No asthma symptoms (Period2; n=70) | 10

ADVERSE EVENTS:
Arm/Group | AZD5069
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD5069 (N=5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstructive airways (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2
Toothache (Gastrointestinal disorders) | 1
Neutropil count decreased (Investigations) | 1
Syncope (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less